CLINICAL TRIAL: NCT05664776
Title: Effect of Dynamic Sitting on Pain Development in Adult Pain Developers in Sedentary Environments - a Randomized Controlled Cross-over Trial
Brief Title: Effect of Dynamic Sitting on Pain Development
Acronym: DynSit-Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Collaborators: Bergardi GmbH (Unknown)
Responsible Party: Principal Investigator, Bernhard Schwartz, Principal Investigator, University of Applied Sciences for Health Professions Upper Austria
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DynSit-Pain
Record Dates: First submitted 2022-12-05; First posted 2022-12-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Lower Back Pain
Keywords: Sedentary Behavior; Occupational Diseases; Pain Developer; Lower Back Pain; Office Environments
MeSH Terms: conditions — Low Back Pain; Sedentary Behavior; Occupational Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (control first) (Experimental): The pre-existing static office chair will be used in the personal workplace for the first 6 weeks within the first half of the study. A wash-out period of a minimum of 4 weeks will be executed after the first half of the study. A dynamic office chair will be used on the personal workstation for 6 weeks within the second half of the study after the wash-out period.
  Interventions: Device: Dynamic office chair
- Arm B (intervention first) (Experimental): A dynamic office chair will be used in the personal workplace for the first 6 weeks within the first half of the study. A wash-out period of a minimum of 4 weeks will be executed after the first half of the study. The pre-existing static office chair will be used on the personal workstation for 6 weeks within the second half of the study after the wash-out period.
  Interventions: Device: Dynamic office chair

INTERVENTIONS:
Device: Dynamic office chair — The dynamic office chair has a typical office chair design (e.g. seat pan and a lumbar support). The seat pan is mounted on a flexible mechanic construction that allows hip movements in the frontal plane while sitting.

SUMMARY:
Worksite based prolonged static sitting postures can cause musculoskeletal pain. While the development of pain increases due to the constant growth of digitalization at work, numerous interventions to reduce prolonged sitting periods have been created. The effects of such interventions have not yet been properly examined. Thus, the "DynSit-Pain" project was initiated to investigate the influence of dynamic sitting on the pain development of pain developers in office environments.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, randomized, controlled, counter-balanced, two-arm field study investigating the effect of dynamic sitting on musculoskeletal pain in office workers classified as pain developers.

The study consists of a pre-screening visit and 4 assessment days / visits. During this pre-screening visit and after proving the study eligibility (inclusion / exclusion criteria), half of the study participants will randomly be allocated to one of the two study arms. Depending on the arm allocation, participants will receive a dynamic (= intervention) or static (= control) office chair for 6 weeks. After a wash-out of at least 4 weeks the 6-week intervention resp. control will be switched. The randomization will be realized with opaque envelopes.

Overall participants will execute the identical assessments within the control and the intervention chair group. The wash-out phase between the control and the intervention periods will ensue identical baseline conditions for both chairs. The overall duration of study participation amounts to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* People aged between 18 and 65 years
* People classified as pain developers (e.g., increase of pain of 10 mm on a 100 mm paper based visual analogue scale) determined by pre-screening
* Office workers
* Employment status: > 30 h / week
* Sufficient German language skills (minimum B2 level)
* Table height of at least 63 cm at the main workplace

Exclusion Criteria:

* Physical or mental limitations that aggravate dynamic sitting or using the interventional chair (e.g., wheel chair users, vestibular dysfunctions)
* Pregnancy
* Working in sitting posture for less than 20 hours per working week in the main workplace.
* Bodyweight over 110 kg and a body height over 195 cm
* Regular therapy or medication for pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Mean change in subjectively perceived lower back pain as determined with a Visual Analogue Scale (VAS) | 6 weeks
  Participants will rate their subjectively perceived lower back pain before and after a conventional occupational day on 5 consecutive days starting at baseline (week 1) and ending with the post-intervention visit (week 6). Subjectively perceived lower back pain will be assessed with a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 points (strongest pain imaginable).
  Question: Please rate the level of your lower back pain at this moment.

SECONDARY OUTCOMES:
Change in impact of pain on daily life (pre- vs. post-intervention) estimated with the German version of the Oswestry Disability Index (ODI-D) | 6 weeks
  Participants will rate their subjectively perceived pain with the German version of the Oswestry Disability Index (ODI-D) at the baseline and post-intervention visits.
  The ODI-D coverts 10 items: Pain intensity, Personal care, Lifting, Walking, Sitting, Standing, Sleeping, Sex (if applicable), Social and Travel. Each item consists of 6 statements which are scored from 0 (lowest disability) to 5 (highest disability).
Mean change in subjectively perceived mental fatigue (pre- vs. post-work, weekly average) estimated via Visual Analogue Scale (VAS) | 6 weeks
  Participants will rate their subjectively perceived mental fatigue before and after a conventional occupational day on 5 consecutive days starting at baseline (week 1) and ending with the post-intervention visit (week 6). Subjectively perceived mental fatigue will be assessed with a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 points (strongest mental fatigue imaginable).
  Question: Please rate the level of your mental fatigue at this moment.
Mean subjectively rated working performance (post-work, weekly average) estimated via VAS | 6 weeks
  Participants will rate their subjectively perceived working performance before and after a conventional occupational day on 5 consecutive days starting at baseline (week 1) and ending with the post-intervention visit (week 6). Subjectively perceived working performance will be assessed with a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (not productive at all) to 100 points (very productive).
  Question: Please rate the level of your working performance on this working day.
Change in quality of life (pre- vs. post-intervention) estimated via 5-level EuroQol quality of life questionnaire (EQ-5D-5L) | 6 weeks
  Participants will rate their subjectively perceived quality of life with the German version of the EQ-5D-5L at the baseline and post-intervention visits.
  The EQ-5D-5L covers 5 Dimensions: Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. Each dimension consists of 5 levels ranging from level 1 (no problems/pain/anxiety) to level 5 (extreme problems/pain/anxiety). It also includes a vertical visual analog scale with a range from 0 (worst imaginable health state) to 100 points (best imaginable health state).
User's experience estimated with the User Experience Questionnaire-Short version (UEQ-S) | 6 weeks
  Subjects will rate the usability of the dynamic chair with the German version of the User Experience Questionnaire-Short version (UEQ-S) at the relevant post-intervention visit.
  The UEQ-S cover both classical usability aspects (efficiency, perspicuity, dependability) and user experience aspects (originality, stimulation). It consists of 8 items, each rated on a seven-point scale with a ranked order. The endpoints of the items are (left to right): obstructive to supportive / complicated to easy / inefficient to efficient / confusing to clear / boring to exciting / not interesting to interesting / conventional to inventive and usual to leading edge.
User's experience via qualitative interview | 6 weeks
  The first five participants using the dynamic chair will be contacted for a qualitative interview regarding the user experience and usability of dynamic sitting. This interview will last for about 60 minutes. After five interviews the data will be analyzed, and the collection will be ceased if data saturation is reached, or else the other 5 participants will be interviewed as well.
Number of adverse events (AE) estimated via an adverse event form sheet | 16 weeks
  In the diary and at all study visits participants will be asked for new adverse events.
Sitting behaviors estimated via microcontrollers | During the 6 weeks of the period of intervention
  The usage of the interventional chair will be tracked (i.e., the system cannot detect which person is sitting on it) by means of a microcontroller to determine if the dynamic chair was used or replaced within the interventional period.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwartz, Dr. BSc MSc, Principal Investigator — FH Gesundheitsberufe OÖ
Locations (1):
- University of Applied Sciences for Health Professions Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No